CLINICAL TRIAL: NCT07382791
Title: The Analysis of Delayed Gastric Emptying After Pancreatic Surgery
Brief Title: Delayed Gastric Emptying After Pancreatic Surgery
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Clinical Professor, National Taiwan University Hospital
Other Study IDs: 20217135RIND
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Neoplasm
Keywords: Pancreatic surgery, Delayed gastric emptying, Gastrointestinal feeding tube
MeSH Terms: conditions — Pancreatic Neoplasms; Gastroparesis | interventions — Pancreatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pancreatectomy group
  Interventions: Procedure: pancreatectomy

INTERVENTIONS:
Procedure: pancreatectomy — All procedures demanding pancreatic parenchyma transaction

SUMMARY:
Delayed gastric emptying (DGE) is a common complication of pancreatic surgery. Once it occurs, it often affects the patient's postoperative quality of life and may even delay subsequent necessary treatments, such as adjuvant chemotherapy. Therefore, this project aims to retrospectively collect basic data, preoperative and postoperative blood tests (blood cell counts, biochemistry, tumor markers, glucose-related, lipid-related), and preoperative and postoperative imaging examinations (CT, MRI, Ultrasound, PET scan, Endoscopy, etc.) of patients who underwent pancreatic surgery at our hospital. We aim to compare whether surgical methods, the placement of gastrointestinal feeding tubes, lesion margin clearance rates, and postoperative remnant pancreatic volume affect the occurrence of delayed gastric emptying and related quality of life. This analysis is intended to understand and analyze the risk factors for delayed gastric emptying in pancreatic surgery patients, the indications for gastrointestinal feeding tube placement, as well as the management and prognosis of delayed gastric emptying, with the expectation of providing more diverse and specific treatment recommendations for patients with delayed gastric emptying after pancreatic surgery in the future.

Keywords: Pancreatic surgery, Delayed gastric emptying, Gastrointestinal feeding tube III. Background Delayed Gastric Emptying after Pancreatic Surgery Delayed gastric emptying is a common complication of pancreatic surgery. However, once it occurs, it often affects the patient's postoperative quality of life and may even delay subsequent necessary treatments, such as adjuvant chemotherapy.

IV. Objectives To compare whether surgical methods, the placement of gastrointestinal feeding tubes, lesion margin clearance rates, and postoperative remnant pancreatic volume affect the occurrence of delayed gastric emptying and related quality of life in patients.

V. Methodology and Procedures Data Collection The Principal Investigator and Co-Investigator will retrospectively collect basic data of patients who underwent pancreatic surgery at this hospital. This includes preoperative and postoperative blood tests (blood counts, biochemistry, tumor markers, glucose-related, lipid-related) and imaging examinations (CT, MRI, Ultrasound, PET scan, Endoscopy, etc.). This data will be used to compare the impact of surgical methods, gastrointestinal feeding tube placement, margin clearance, and remnant pancreatic volume on the occurrence of delayed gastric emptying and related quality of life. The goal is to understand and analyze risk factors, indications for feeding tube placement, management, and prognosis.

From the hospital portal system, approximately 500 medical records of patients with pancreatic diseases who underwent pancreatic surgery or invasive treatment performed by the Principal Investigator and Co-Investigator between January 2005 and July 2021 will be collected. This observational study will collect routine imaging and laboratory tests performed at the hospital to analyze treatment indications, surgical indicators, and prognosis.

Inclusion Criteria:

1. Males or females aged 20 years or older.
2. Patients scheduled to undergo pancreatic surgery.

Exclusion Criteria:

1. Patients under 20 years of age at this hospital.
2. Presence of other active malignancies prior to diagnosis.
3. Minors, pregnant women, breastfeeding women, and patients with psychiatric disorders.

Statistical Analysis Patient medical records will be utilized to analyze risk factors for delayed gastric emptying, indications for gastrointestinal feeding tube placement, management, and prognosis for patients undergoing pancreatic surgery, aiming to provide diverse and specific treatment recommendations in the future.

Confidentiality and Privacy Protection To ensure patient privacy and personal information security, after querying the relevant data of enrolled subjects, the data sheet will use new codes to represent the subjects' identities. Experimenters and analysts will only have access to this de-linked data sheet for analysis. All electronic data will be password-protected and accessible only by specific personnel related to this project.

All data not used or after analysis will be stored at the NTU Department of Surgery for 15 years and then destroyed by shredder or incineration to remove identifiable personal data, unless required for medical or research purposes. Researchers (including external personnel) will sign a written pledge stating that medical record data will not be reused, disclosed to third parties, or used for purposes outside this study, unless required by law or audited by the Research Ethics Committee.

Budget and Equipment Item Purpose Amount (TWD) Database Analysis Software Data Analysis 50,000 Statistical Consulting Data Analysis 50,000 Statistical Consulting Chart Creation 50,000 English Editing, Publication, Printing, Stationery Thesis Publication 50,000 Part-time Student

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 20 years or older.
2. Patients scheduled to undergo pancreatic surgery.

Exclusion Criteria:

1. Patients under 20 years of age at this hospital.
2. Presence of other active malignancies prior to diagnosis.
3. Minors, pregnant women, breastfeeding women, and patients with psychiatric disorders.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients received pancreatectomy at National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of nasogastric tube intubation after surgery | 3 months after poancreatetcomy

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwn, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided